CLINICAL TRIAL: NCT04690569
Title: Prospective, Multi-Center, Observational, Blinded Study to Establish the Diagnostic Performance of the MeMed BV™ Test for Differentiating Bacterial From Viral Infection in Patients With Suspected Acute Bacterial or Viral Infection ("APOLLO" STUDY)
Brief Title: Establish MeMed BV™ Performance for Differentiating Bacterial From Viral Infection in Suspected Acute Infection Patients (APOLLO STUDY)
Acronym: Apollo
Status: Completed | Type: Observational
Sponsor: MeMed Diagnostics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MMD010
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Acute Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Infectious: Eligible pediatric and adult patients from ED\Urgent care and hospital admitted, with symptoms consistent with acute bacterial or viral infection.
  Interventions: Diagnostic Test: MeMed BV
- Healthy: For the purpose of establishing a normal reference range.
  Interventions: Diagnostic Test: MeMed BV

INTERVENTIONS:
Diagnostic Test: MeMed BV — The MeMed BV™ Test is an immunoassay that measures three non-microbial (host) proteins (TRAIL, IP-10, and CRP) in adult and pediatric serum samples. The test is intended for use in conjunction with clinical assessments and other laboratory findings as an aid to differentiate bacterial from viral infection. The test is indicated for use in patients presenting to the ED, urgent care center and inpatients with suspected acute bacterial or viral infection. The MeMed BV™ Test generates a numeric score that falls within discrete interpretation bins based on the increasing likelihood of bacterial infection. The MeMed BV™ test is intended for in vitro diagnostic use only.

SUMMARY:
Prospective, multi-center, observational, blinded study, enrolling pediatric and adult subjects. Eligible ED\Urgent care and hospital admitted patients with symptoms consistent with acute bacterial or viral infection and healthy subjects will be recruited according to the eligibility criteria. Each participant will undergo a thorough investigation upon recruitment that includes documenting clinical, radiological, laboratory and microbiological information for determining their health status.

Follow-up data will be collected via a phone call. Diagnostic performance of the MeMed BV™ Test for differentiating bacterial from viral infection will be assessed using an expert adjudication comparator method.

The study will be run in a blinded fashion: site personnel will be blinded to the comparator method outcomes, and the expert panel will be blinded to the results of the index test. Results of the index test will not be revealed to the attending clinician and so will not influence patient management.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained from the patient or his/her legal guardian. For children under 18 years old, written informed consent from the legal guardian and assent from the patient (depending on the local requirements)
* Over 90 days of age
* Clinical suspicion of acute bacterial or viral infection
* Temperature ≥ 37.8°C (100°F) (any body site, any measurement device, including self-reported) or tactile fever, either of them noted at least once within the last 7 days
* Current disease duration ≤ 7 days

Exclusion Criteria:

* Another unrelated episode of febrile infection within the past 2 weeks
* Suspicion and/or confirmed diagnosis of infectious gastroenteritis/ colitis
* >48 hours of oral antibiotic treatment
* >12 hours of intravenous\intramuscular antibiotic treatment
* HIV, HBV, or HCV infection (self-declared or known from medical records)
* A proven or suspected infection on presentation with Mycobacterial (e.g. Tuberculosis, MAC), parasitic or fungal (e.g. Candida, Histoplasma, Aspergillus) pathogen
* Active inflammatory disease (e.g. IBD, SLE, JIA, RA, Kawasaki, other vasculitis)
* Major trauma and\or burns in the last 7 days
* Major surgery in the last 7 days
* Congenital immune deficiency (CID)
* Acquired immune deficiency\modulation state including:

  * Active malignancy
  * Current treatment with immune-suppressive or immune-modulating therapies, including without limitations:

    * Administration of P.O.\IV\IM high dose steroids >1mg/kg/day prednisone (or equivalent) at some point in the past 10 days or daily continuous use of steroids > 0.25 mg/kg/day in the past 7 days
    * Monoclonal antibodies, anti-TNF agents
    * Intravenous immunoglobulin (IVIG)
    * Cyclosporine, Cyclophosphamide, Tacrolimus, Azathioprine, Methotrexate
    * G/GM-CSF, Interferons
  * Post solid organ/bone marrow transplant patients
  * Asplenia, sickle cell disease
* Indwelling central venous catheter
* Cystic Fibrosis
* Pregnancy- self reported or medically known
* Other severe illnesses that affect life expectancy and quality of life such as:

  * Severe psychomotor retardation
  * Congenital metabolic disorder
  * End stage renal disease, advanced heart failure (NYHA 3/4), advanced COPD (GOLD 3/4)

Min Age: 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospital admitted, ED and urgent care center patients over the age of 90 days, with suspected acute bacterial or viral infection and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1384 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-11-22 (Actual); Study Completion 2020-11-22 (Actual)

PRIMARY OUTCOMES:
Establish the diagnostic performance of the MeMed BV™ Test for differentiating bacterial from viral infection using expert adjudication comparator method. | Through study completion, an average of 18 months
  Establish the diagnostic performance of the MeMed BV™ Test for differentiating bacterial from viral infection using expert adjudication comparator method.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - Johns Hopkins, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Maimonides Medical Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - American Family Care Urgent Care, Easley, South Carolina
  - American Family Care Urgent Care, Powdersville, South Carolina
  - American Family Care Urgent Care, Chattanooga, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas
- Israel (2):
  - Hillel Yaffe Medical Center, Hadera
  - Carmel Medical Center, Haifa